CLINICAL TRIAL: NCT05844605
Title: Joan Ribas Araquistain Program for Research and Therapeutic Innovation in Prehabilitation, Rehabilitation and Comprehensive Approach to the Sequelae of Brain Tumors
Brief Title: Prehabilitation, Rehabilitation and Comprehensive Approach to the Sequelae of Brain Tumors
Acronym: PREHABILITA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Guttmann (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020330
Record Dates: First submitted 2023-03-10; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Brain Tumor
Keywords: brain tumour; prehabilitation; neuromodulation; motor training; cognitive training
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Pilot single-cohort feasibility open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation (Experimental): Adult patients affected by Brain Tumour and candidated for surgical treatment.
  Interventions: Procedure: Non-invasive neuromodulation (TMS and/or tDCS)

INTERVENTIONS:
Procedure: Non-invasive neuromodulation (TMS and/or tDCS) — Non-invasive neuromodulation (TMS and/or tDCS) coupled with intensive behavioural training (neurorehabilitation and/or cognitive rehabilitation)

SUMMARY:
The goal of the present pilot single-cohort feasibility trial is to investigate the feasibility and understand potential mechanisms of efficacy for Neuromodulation-Induced Cortical Prehabilitation (NICP) in adults with brain tumours and eligible for neurosurgery.

The main questions it aims to answer are:

* is the intervention feasible, in terms of adherence, retention, safety and patient's satisfaction;
* what are the mechanisms of neuroplasticity primed by NICP

Participants will undergo a prehabilitation protocol, consisting of daily sessions (total: 10-20 sessions) structured as follows:

* Intervention 1: non-invasive neuromodulation (TMS/tDCS).
* Intervention 2: motor and/or cognitive training, during or immediately after non-invasive neuromodulation, for about 60 minutes.

The timeline is structured as follows:

T1: baseline (before NICP) T2-T3: NICP period T4: after NICP T5: surgery T6: after surgery

Clinical, neuroimaging and neurophysiology assessments will be performed before NICP (T1), after NICP (T4), and after neurosurgery (T6). Feasibility outcomes will be determined during NICP protocol (T2-T3).

The objective of the proposed intervention is to progressively reduce the functional relevance of eloquent areas, which are healthy brain areas close with the tumour and thus exposed to the risk of being lesioned during surgery. In fact, previous studies have shown that temporary inhibition of eloquent areas (by neuromodulation) coupled with intensive motor/cognitive training promoted the activation of alternative brain resources, with a shift of functional activity from eloquent areas to areas functionally related, but anatomically distant from the tumour.

By moving the activation of key motor/cognitive functions away from the tumour, the risk of postoperative functional sequelae will be reduced; which in turn will falicitate a more radical tumour excision by the neurosurgeon.

DETAILED DESCRIPTION:
Neuromodulation-Induced Cortical Prehabilitation (NICP) is a relatively new approach in the neurosurgical field. It consists of priming neuroplastic changes before neurosurgery for brain tumours, in order to improve surgical outcomes and, hopefully, long-term survival and quality of life. The intervention comprises two elements:

1. Neuromodulation (like transcranial magnetic stimulation, TMS, and transcranial direct current stimulation, tDCS). The goal of neuromodulation is to inhibit the eloquent areas, defined as brain areas functionally active and close to the tumour.
2. Behavioural training (like motor training, cognitive training, or a combination). The function trained corresponds with the function of the eloquent area targeted by neuromodulation.

The two interventions are provided on a daily basis, and repeated over 10-20 consecutive weekdays. Notably, after the inhibition of the eloquent area there is a temporal window of about one hour, where intensive training of the same function requires the activation of alternative areas/pathways. By consolidating this alternative activation over multiple sessions, the outcome is a reduction in the functional relevance of eloquent areas, in favour of alternative resources anatomically distant from the tumour.

Only few case reports have been published so far, with very positive results obtained by means of invasive neuromodulation; the term 'invasive' means that a first neurosurgery was required to implant electrodes over eloquent areas for intracranial electrical stimulation, followed after few days/weeks by a second surgery for tumour removal. Despite relevant neuroplastic changes, the problem with this approach has been the high rate of adverse events occurred (infections, edema, pain, seizure) due to the invasiveness of the procedures. Therefore, by using a non-invasive neuromodulation approach, the goal of the present trial is to promote neuroplastic changes beneficial for neurosurgery, while at the same time ensuring no serious adverse events.

Further details on neuromodulation. Investigators will apply the most appropriate neuromodulation protocol, personalized based on whether to perform TMS and/or tDCS, individual resting motor threshold (for TMS), and target determination (related to eloquent areas).

Protocol for low frequency rTMS:

* intensity: 90% RMT;
* frequency: 1 Hertz;
* total number of pulses: 1600.

Protocol for tDCS:

* cathode: over eloquent areas
* anode: typically over areas that should be activated, as opposed to eloquent areas

Further details on upper limb prehabilitation training.

Within the 60 minutes immediately after neuromodulation, patients will perform an intensive training of the same function of the eloquent area, which is now temporarily inhibited. Intensity of the training will be continuously adjusted in terms of type, difficulty and variability:

* Type: exercises specific for finger individuation (play the piano, typewriting), finger coordination (dexterity, manipulation), arm reaching. In order to integrate upper limb function with other motor-cognitive functions, dual task training will be performed, both motor-cognitive (decision making, stroop task, motor sequence learning etc.) and motor-motor (bimanual activites, arm and balance tasks, etc.);
* Difficulty: the intensity of the exercise will be set as to result 'difficult, yet achievable' by the patient. This way it is ensured that the brain is under a stress condition which, together with concurrent eloquent area inhibition, will promote and consolidate the activation of alternative resources.
* Variability: varying systematically the type and difficulty of the training is useful to keep the patient engaged and ensure that the end result will be a global motor-cognitive training, instead of a monotonic improvement in a specific performance.

Further details on Prehabilitation for language and cognitive training. Language-cognitive training will follow the same rationale illustrated for motor training. Soon after neuromodulation the patient will perform a computerized cognitive training on a dedicated platform ("Guttmann NeuroPersonalTrainer"® (GNPT). Exercises will be customized based on specific patient's deficits, and/or functions at risk of being compromised after surgery. For instance, the neuropsychologist may vary settings such as presentation speed, latency time or number of images, thus finely tuning several difficulty levels. Regarding language, tasks will be planned and supervised in a personalized way by a neuropsychologist, readjusting their planning if necessary.

Discontinuation, adherence, and permission for concomitant care.

The intervention will be discontinued in the following cases:

* participant's request;
* serious adverse events attributable to the intervention. Patients will be allowed to continue any ongoing treatment. Formal training of motor-cognitive functions outside the protocol will be discourage, as it may affect neuroplastic changes in an unpredictable way.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of brain tumour requiring neurosurgery
* ability to undertake at least 10 sessions of prehabilitation protocol
* tumour location posing the patient at risk of developing post-operative neurological deficits, for instance at the level of upper limb motor function and speech production
* ability to understand the general purpose of the prehabilitation program and understand simple instructions
* being willing to participate and sign the informed consent
* being able to sit unassisted for one hour.

Exclusion Criteria:

* any contraindication for magnetic resonance imaging or transcranial magnetic stimulation
* unstable medical conditions
* musculoskeletal disorders that may significantly affect functional training
* pain, depression, fatigue that may significantly affect functional training
* history of alcohol/drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility_adherence | Throughout the intervention, which will last approximately 10 to 20 sessions (two to four weeks)
  Sufficient adherence is defined by attending at least 75% of the planned sessions
Feasibility_retention | Throughout the intervention, which will last approximately 10 to 20 sessions (two to four weeks)
  Sufficient retention is defined by at least 75% of enrolled patients completing the intervention
Feasibility_safety | Throughout the intervention, which will last approximately 10 to 20 sessions (two to four weeks)
  Adequate safety is defined by the absence of any serious adverse event
Feasibility_patient's satisfaction | Throughout the intervention, which will last approximately 10 to 20 sessions (two to four weeks)
  Self reported patient's satisfaction, as from the EORTC* PATSAT C-33 questionnaire.
  All of the EORTC scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. in this case, higher score means higher patient's satisaction of the treatment received.
  *European Organisation for Research and Treatment of Cancer (EORTC)

SECONDARY OUTCOMES:
Clinical_Neurological Assessment in Neuro-Oncology (NANO) scale | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Standardized assessment of neurological functional status in patients with brain tumour.
  Score ranges from 0 to 27, with higher scores indicating worse neurological status.
Clinical_Karnofsky Performance Status | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of functional independency for patients with brain tumour. Score ranges from 0 to 100, with higher scores representing higher levels of functional independency.
Clinical_upper limb_9 Hole Peg Test | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of hand dexterity. Results are measured in seconds to complete a dexterity task (take pegs one at a time from a container and place in nine holes, and then back in the container). The lower the time taken to complete the task, the better the performance.
Clinical_upperl limb_Fugl-Meyer Upper Extremity | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of upper limb motor impairment. Score ranges from 0 to 66, with higher scores indicating better motor function.
Clinical_upper limb_Hand dynamometer | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of grip strength. Results are measured in kg, with higher scores indicating higher grip strength.
Clinical_upper limb_Deary-Liewald reaction time task | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Computerized assessment of efficiency of basic processes for perception and response execution. Results are measured as time (milliseconds) between stimulus presentation and response execution. The shorter the time interval, the better the performance.
Clinical_lower limb and balance_Fugl Meyer Lower Extremity | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of lower limb motor impairment. Score ranges from 0 to 34, with higher scores indicating better motor function.
Clinical_lower limb and balance_Brunel Balance Assessment | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of balance. Score ranges from 0 to 12, with higher scores indicating better performance.
Clinical_lower limb and balance_Six minute walking test | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Submaximal test of aerobic capacity. Results are measured as the total distance (meters) walked during six minutes. The longer the distance, the better the performance.
Clinical_EORTC-QLQ-C30* | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  questionnaire of quality of life for oncological patients. All of the EORTC scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status represents a high quality of life, but a high score for a symptom scale represents a high level of symptomatology / problems.
  *European Organisation for Research and Treatment of Cancer (EORTC) QLQ: quality of life questionnaire
Clinical_EORTC-BN20 | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  EORTC* brain cancer module. All of the EORTC scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. In this case, a high score for a symptom scale represents a high level of symptomatology / problems.
  *European Organisation for Research and Treatment of Cancer (EORTC)
Clinical_EORTC-FA12 | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  EORTC* fatigue module. All of the EORTC scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. In this case, a high score for a symptom scale represents a high level of fatigue.
  *European Organisation for Research and Treatment of Cancer (EORTC)
Clinical_Revised Barcelona Test | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Battery of clinical assessments for high cognitive functions, including: language, writing, reading, memory, imitation of gestures and postures, constructive praxis, orientation, arithmetics and comprehension.
  Normative data indicate a mean of 100 and standard deviations of 15, range 40-160.
  Higher score means better performance. Scores under 80 are considered below the normality.
Clinical_WAIS-III Wechsler Adult Intelligence Scale | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of verbal, manipulative and total intelligent quotient. Normative data indicate a mean of 100 and standard deviations of 15, range 40-160.
  Higher score means better performance. Scores under 80 are considered below the normality.
Clinical_Trail Making Test | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of visual attention, sequencing, flexibility and graphomotor ability.
  Results are reported as time to complete the task, and number of errors. Higher score means worse performance.
Clinical_Continuous Performance Test-III | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of sustained attention. Results are reported as reaction time, and number of errors (omission and commission). Higher score means worse performance.
Clinical_Rey Auditory Verbal Learning Test | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of auditory verbal memory. Score ranges between 0 and 75 (immediate memory), 0 and 15 (delayed memory), 0 and 15 (recognition- errors (commission and ommission). The higher the score, the better the performance.
Clinical_WMS-IV Wechsler Memory Scale | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of memory functions. Normative data indicate a mean of 100 and standard deviations of 15, range 40-160.
  Higher score means better performance. Scores under 80 are considered below the normality.
Clinical_Symbol Digit Modalities Test | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of visual tracking, concentration and visuomotor speed. Total score is the result of summing the number of correct substitutions within the 90 second interval (max = 110). Higher score means better performance.
Clinical_PMR Verbal fluency by letters. | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of lexical access and verbal fluency. Count up the total number of words beginning with the requested letter that the person is able to produce in one minute. Three letters (PMR) are requested and the final score is the sum of the three attempts. Higher scores means better performance.
Clinical_Hayling Test | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of behavioural regulation, initiation speed and response inhibition. The test is divided in part A (0-15) and B (0-45). Answers are classified as correct (0 points) or incorrect (1 point) and reaction time is also measured. Higher score (more errors) imply a lower performance.
Clinical_Wisconsin Card Sorting Test | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of executive function. Outcome measures of categories achieved (higher means better performance), trials, errors, and perseverative errors (the lower the score, the greater the efficiency of the examinee in the task)
Clinical_Hospital Anxiety and Depression Scale | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Clinical assessment of anxiety and depression. The total score is the sum of each item. Final score ranges from 0 to 21 with the highest scores indicating the highest levels of anxiety and depression: 0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe).
Neuroimaging_structural MRI | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Assessment of tumour location, volume (voxels, cm3) and distribution (based on neuroanatomical atlases)
Neuroimaging_resting state fMRI | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Assessment of regional interaction in the brain (Blood-oxygen-level-dependent contrast imaging), during a rest condition.
  High resolution multiband (anterior posterior phase-encoding, acceleration factor = 8) interleaved acquisitions (T2 - weighted echo-planar imaging scans, repetition time = 800 ms, echo time = 37 ms, 750 volumes, 72 slices, slice thickness = 2 mm, Field-of-view = 208 mm).
Neuroimaging_fMRI_Word generation task | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Assessment of brain activity (Blood-oxygen-level-dependent contrast imaging) when the patient is asked to mention words starting with a certain letter.
  High resolution multiband (anterior posterior phase-encoding, acceleration factor = 8) interleaved acquisitions (T2 - weighted echo-planar imaging scans, repetition time = 800 ms, echo time = 37 ms, 750 volumes, 72 slices, slice thickness = 2 mm, Field-of-view = 208 mm).
Neuroimaging_fMRI_Semantic decision task | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Assessment of brain activity (Blood-oxygen-level-dependent contrast imaging) when the patient is asked to mention objects from certain places.
  High resolution multiband (anterior posterior phase-encoding, acceleration factor = 8) interleaved acquisitions (T2 - weighted echo-planar imaging scans, repetition time = 800 ms, echo time = 37 ms, 750 volumes, 72 slices, slice thickness = 2 mm, Field-of-view = 208 mm).
Neuroimaging_fMRI_Comprehensive auditive task | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Assessment of brain activity (Blood-oxygen-level-dependent contrast imaging) when the patient is asked to listen to a story.
  High resolution multiband (anterior posterior phase-encoding, acceleration factor = 8) interleaved acquisitions (T2 - weighted echo-planar imaging scans, repetition time = 800 ms, echo time = 37 ms, 750 volumes, 72 slices, slice thickness = 2 mm, Field-of-view = 208 mm).
Neuroimaging_fMRI_Finger tapping task | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Assessment of brain activity (Blood-oxygen-level-dependent contrast imaging) when the patient is asked to perform a fingering exercise.
  High resolution multiband (anterior posterior phase-encoding, acceleration factor = 8) interleaved acquisitions (T2 - weighted echo-planar imaging scans, repetition time = 800 ms, echo time = 37 ms, 750 volumes, 72 slices, slice thickness = 2 mm, Field-of-view = 208 mm).
Neuroimaging_fMRI_Ankle flexion task | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Assessment of brain activity (Blood-oxygen-level-dependent contrast imaging) when the patient is asked to move the corresponding foot up and down slowly.
  High resolution multiband (anterior posterior phase-encoding, acceleration factor = 8) interleaved acquisitions (T2 - weighted echo-planar imaging scans, repetition time = 800 ms, echo time = 37 ms, 750 volumes, 72 slices, slice thickness = 2 mm, Field-of-view = 208 mm).
Neuroimaging_fMRI_Tongue movement task | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Assessment of brain activity (Blood-oxygen-level-dependent contrast imaging) when the patient is asked to move the tongue in circles, without opening the mouth.
  High resolution multiband (anterior posterior phase-encoding, acceleration factor = 8) interleaved acquisitions (T2 - weighted echo-planar imaging scans, repetition time = 800 ms, echo time = 37 ms, 750 volumes, 72 slices, slice thickness = 2 mm, Field-of-view = 208 mm).
Neurophysiology_TMS mapping_hotspot | Baseline (before the intervention protocol)
  Determination of the cortical target (x, y, z coordinates ijn MNI space) where motor evoked potentials were elicited with the lowest TMS stimulus intensity.
  The muscle used as reference is the first dorsal interosseus (electrodes placed with belly-tendon montage).
  Motor evoked potentials (MEP) are defined as those voltages produced 25 to 50 milliseconds after the TMS stimulus, with a peak-to-peak amplitude of at least 50 microVolts.
Neurophysiology_TMS mapping_resting motor threshold | Baseline (before the intervention protocol)
  Determination of the resting motor threshold (RMT), relatively to the hotspot. A cortical target is defined as MEP positive if at least 3 out of 6 MEP could be elicited.
  To determine RMT, stimulus intensity is progressively reduced until less than 3 MEP out of 6 are elicited. RMT corresponds to this stimulus intensity + 1.
Neurophysiology_TMS mapping_motor function | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Mapping of the motor area for the first dorsal interosseus, with intensity of 120% RMT.
  5 stimuli are delivered to each cortical target, with 5 seconds of interval in between. Cortical mapping is then created by averaging the peak-to-peak amplitude (microVolts) resulting from the stimulation of each target.
Neurophysiology_TMS mapping_language function | At baseline (before the intervention), at the end of the intervention (but before neurosurgery), and at the first available follow up (from one month up to one year after surgery)
  Mapping of language function in regions corresponding to Broca and Wernicke areas, with intensity of 90% RMT (one train of 5 pulses, 5 Hertz). Images are presented, one at a time, on a screen placed in front of the patient. At the same of image presentation, stimulation is delivered (for a total of one second), and audio recording initiates (for a total of 4 seconds). A neuropsychologist is present to determine whether there was any interference in the verbal response due to TMS stimulation.
  If any interference appears, for instance paraphasia o anomia, the cortical target is considered positive for language, hence functionally related to speech processing; otherwise, it is considered negative.
Surgical outcomes | Within the first week after surgery
  Descriptive report of surgical outcomes, including results from intraoperative brain mapping, the absolute and relative volume (voxels, cm3) of tumour removed, adverse events, neurological status post-surgery, and tumour classification based on clinical and histological findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Guttmann, Badalona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study will be available from the corresponding author, upon reasonable request. Alternatively, an online data repository named "Joan Ribas Araquistain Dataset on BRAIN TUMOR PREHABILITATION" will be created and made accessible upon reasonable request to accredited clinicians, researchers, and institutions in the field of neuro-oncology. Furthermore, will sought to establish collaboration agreements with international oncology databases, such as the Georgetown Database of Cancer (G-DOC), REMBRANDT (REpository for Molecular BRAin Neoplasia DaTA) and the Cancer Imaging Archive.

REFERENCES:
- [Background] Duffau H. Lessons from brain mapping in surgery for low-grade glioma: insights into associations between tumour and brain plasticity. Lancet Neurol. 2005 Aug;4(8):476-86. doi: 10.1016/S1474-4422(05)70140-X. PMID 16033690
- [Background] Rivera-Rivera PA, Rios-Lago M, Sanchez-Casarrubios S, Salazar O, Yus M, Gonzalez-Hidalgo M, Sanz A, Avecillas-Chasin J, Alvarez-Linera J, Pascual-Leone A, Oliviero A, Barcia JA. Cortical plasticity catalyzed by prehabilitation enables extensive resection of brain tumors in eloquent areas. J Neurosurg. 2017 Apr;126(4):1323-1333. doi: 10.3171/2016.2.JNS152485. Epub 2016 May 20. PMID 27203145
- [Background] Duffau H. Can Non-invasive Brain Stimulation Be Considered to Facilitate Reoperation for Low-Grade Glioma Relapse by Eliciting Neuroplasticity? Front Neurol. 2020 Nov 12;11:582489. doi: 10.3389/fneur.2020.582489. eCollection 2020. No abstract available. PMID 33304307
- [Background] Hamer RP, Yeo TT. Current Status of Neuromodulation-Induced Cortical Prehabilitation and Considerations for Treatment Pathways in Lower-Grade Glioma Surgery. Life (Basel). 2022 Mar 22;12(4):466. doi: 10.3390/life12040466. PMID 35454957
- [Background] Barcia JA, Sanz A, Gonzalez-Hidalgo M, de Las Heras C, Alonso-Lera P, Diaz P, Pascual-Leone A, Oliviero A, Ortiz T. rTMS stimulation to induce plastic changes at the language motor area in a patient with a left recidivant brain tumor affecting Broca's area. Neurocase. 2012;18(2):132-8. doi: 10.1080/13554794.2011.568500. Epub 2011 Jul 25. PMID 21780986
- [Background] Barcia JA, Sanz A, Balugo P, Alonso-Lera P, Brin JR, Yus M, Gonzalez-Hidalgo M, Acedo VM, Oliviero A. High-frequency cortical subdural stimulation enhanced plasticity in surgery of a tumor in Broca's area. Neuroreport. 2012 Mar 28;23(5):304-9. doi: 10.1097/WNR.0b013e3283513307. PMID 22336871
- [Background] Serrano-Castro PJ, Ros-Lopez B, Fernandez-Sanchez VE, Garcia-Casares N, Munoz-Becerra L, Cabezudo-Garcia P, Aguilar-Castillo MJ, Vidal-Denis M, Cruz-Andreotti E, Postigo-Pozo MJ, Estivill-Torrus G, Ibanez-Botella G. Neuroplasticity and Epilepsy Surgery in Brain Eloquent Areas: Case Report. Front Neurol. 2020 Jul 29;11:698. doi: 10.3389/fneur.2020.00698. eCollection 2020. PMID 32849188
- [Background] Hoogendam JM, Ramakers GM, Di Lazzaro V. Physiology of repetitive transcranial magnetic stimulation of the human brain. Brain Stimul. 2010 Apr;3(2):95-118. doi: 10.1016/j.brs.2009.10.005. Epub 2009 Nov 24. PMID 20633438
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Derived] Boccuni L, Abellaneda-Perez K, Martin-Fernandez J, Leno-Colorado D, Roca-Ventura A, Prats Bisbe A, Buloz-Osorio EA, Bartres-Faz D, Bargallo N, Cabello-Toscano M, Pariente JC, Munoz-Moreno E, Trompetto C, Marinelli L, Villalba-Martinez G, Duffau H, Pascual-Leone A, Tormos Munoz JM. Neuromodulation-induced prehabilitation to leverage neuroplasticity before brain tumor surgery: a single-cohort feasibility trial protocol. Front Neurol. 2023 Oct 2;14:1243857. doi: 10.3389/fneur.2023.1243857. eCollection 2023. PMID 37849833
- See also: webpage of the project — https://www.guttmann.com/en/prehabilita-project